CLINICAL TRIAL: NCT01841606
Title: The Effect of Ondansetron on Cardiac Output in Elective Cesarean Deliveries Under Spinal Anesthesia: A Randomized Controlled Trial
Brief Title: The Effect of Ondansetron on Cardiac Output in Elective Cesarean Deliveries
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Vit Gunka, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H12-03634
Record Dates: First submitted 2013-03-11; First posted 2013-04-26 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Cardiac Output
Keywords: Spinal anesthesia; Elective cesarean deliveries; Ondansetron
MeSH Terms: interventions — Ondansetron; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ondansetron (Experimental): 4mg of IV ondansetron 5 minutes prior to initiation of spinal anesthesia
  Interventions: Drug: Ondansetron
- Placebo (Placebo Comparator): 10mL of IV normal saline 5 minutes prior to initiation of spinal anesthesia
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Ondansetron — 4mg of IV ondansetron
  Other Names: Zofran
  Arms: Ondansetron
Other: Normal saline — 10mL of IV normal saline
  Arms: Placebo

SUMMARY:
Ondansetron is a medication routinely given to mothers having cesarean deliveries to help prevent and treat nausea and vomiting. The investigators are studying the hemodynamic effects of prophylactic ondansetron on parturients undergoing elective cesarean deliveries under spinal anesthesia.

DETAILED DESCRIPTION:
Spinal anesthesia is a routine anesthetic technique for elective cesarean deliveries. Although this provides safe and effective surgical anesthesia, it is not without side effects, including both hypotension and bradycardia. The incidence of hypotension following spinal anesthesia has been estimated to be as high as 80% in an obstetric population. A number of factors are also likely involved in the development of hypotension and bradycardia, including the Bezold-Jarisch Reflex (BJR).

Two human studies with spinal anesthesia, one in an obstetric population, have demonstrated ondansetron's ability to presumably attenuate the BJR and better prevent hypotension by antagonism of 5-HT3 receptors. Maintenance of blood pressure and heart rate are vitally important, as they are required for adequate perfusion of the fetus prior to delivery.

The investigators plan to investigate the hemodynamic effects of prophylactic ondansetron on parturients undergoing elective cesarean deliveries under spinal anesthesia.

Ondansetron is classified as a Pregnancy Category B drug by the FDA, meaning that no adverse fetal effects have been demonstrated in animal studies, but that there is a lack of well controlled studies in pregnant humans.

ELIGIBILITY:
Inclusion Criteria:

* Elective CD under spinal anesthesia
* Fluency in English

Exclusion Criteria:

* Contraindication to spinal anesthesiA
* Allergy to ondansetron

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vit Gunka, MD FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Ondansetron: Patients receiving pre-spinal ondansetron
- Placebo: Patients receiving placebo
Period: Overall Study
Arm/Group | Ondansetron | Placebo
Started | 25 | 27
Completed | 25 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ondansetron: 4mg IV Ondansetron
- Placebo: 10mL IV normal saline
- Total: Total of all reporting groups
Arm/Group | Ondansetron | Placebo | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.32 (3.86) | 34.7 (4.76) | 34.5 (4.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 52
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 25 | 27 | 52

OUTCOME MEASURES:

1. Primary Outcome: Change in Cardiac Output From Baseline to 20 Minutes Post-spinal
Description: Maximum change in cardiac output from initiation of spinal anesthesia (baseline) until uterine incision (20 minutes post-spinal)
Time Frame: Baseline and 20 minutes
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Ondansetron | Placebo
Number analyzed (Participants) | 25 | 27
L/min | -2.05 (1.43) | -1.92 (1.41)

ADVERSE EVENTS:
Arm/Group | Ondansetron | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 0/25 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No